CLINICAL TRIAL: NCT04714138
Title: Remote Evaluation of Quality of Life and Functional Capacities in Patients Hospitalised for COVID-19: a Prospective Observational Study
Brief Title: Remote Video Consultation for Quality of Life Assessment in Patients Hospitalised After COVID-19 Infection
Acronym: TELECOVID
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier du Havre (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A03110-39
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Around 90.000 patients have been hospitalised due to COVID-19 infection in France between March 1st and June 15th; 19% of those requiring intensive care. Approximately 80% of these patients have been discharged home by September 30th. Nonetheless, COVID-19 infection along with intensive care consequences are very likely to impede those patients quality of life and functional capacities.

This study aims to describe the quality of life outcomes and functional capacities of COVID-19 survivors, at least 6 months after primary care hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* COVID-19 hospitalisation at Le Havre hospital between March 1st and May 11th
* Non-opposition during first phone contact

Exclusion Criteria:

* Guardianship
* Juvenile patients
* Pregnancy
* Inability to communicate
* Cognitive disorders
* Deceased patient

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COVID-19 adults patients hospitalised at Le Havre hospital between March 1st and May 11th
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | 10 to 12 months after hospital discharge during remote video consultation
  Measured with the Short-Form health survey (SF-36) scale (score ranging form 0 (worst score) to 100 (best score) per item)

SECONDARY OUTCOMES:
Functional capacity | 10 to 12 months after hospital discharge during remote video consultation
  One-minute Sit-to-stand test
Independency | 10 to 12 months after hospital discharge during remote video consultation
  KATZ score (ranging 0 (fully dependent) to 6 (fully independent))

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Du Havre, Montivilliers, Normandy, France

IPD SHARING:
Plan to Share IPD: Undecided